CLINICAL TRIAL: NCT03310892
Title: Patient-directed Messaging to Increase Colorectal Cancer Screening
Brief Title: Tailored Messaging for CRC Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 827866
Record Dates: First submitted 2017-10-05; First posted 2017-10-16 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Participants in this arm will Usual scheduling process without any intervention
- Generic Message (Experimental): Participants in this arm will receive a telephone call from a study team member, and if no answer, up to two additional attempts will be made. During the telephone call, the study team member will ask the participant a series of 7 questions then receive a "generic" message encouraging colonoscopy scheduling.
  Interventions: Behavioral: Generic message
- Tailored Message (Experimental): Participants in this arm will receive a telephone call from a study team member, and if no answer, up to two additional attempts will be made. During the telephone call, the participant will answer a series of 7 questions then receive a "tailored" message encouraging colonoscopy scheduling, which will be determined by their responses to the preceding questions.
  Interventions: Behavioral: Tailored message

INTERVENTIONS:
Behavioral: Generic message — Generic message
  Arms: Generic Message
Behavioral: Tailored message — Tailored message
  Arms: Tailored Message

SUMMARY:
This is a randomized controlled trial to to determine whether direct, tailored messaging to patients prior to scheduling colonoscopy will increase patient adherence to provider recommendation for screening colonoscopy.

DETAILED DESCRIPTION:
The proposed study is a prospective, randomized trial. All eligible subjects (patients identified to be contacted to schedule screening colonoscopy) will be randomized to one of three study arms: usual scheduling process (control), a generic message arm, or a tailored message arm. Patients in the "tailored message" arm will receive a telephone call and be asked a series of questions that will be used to assign patients to one of four messaging cohorts. After these questions have been answered, the patient will then receive a tailored message corresponding to his or her respective messaging cohort, encouraging them to schedule a colonoscopy with a directed script. In the "generic message" arm, patients will receive a telephone call and be asked to answer the same series of questions as the "tailored message" group, then receive a single, standard script encouraging them to schedule a colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. University of Pennsylvania Health System (UPHS) patients with an active order for screening or surveillance colonoscopy without an existing colonoscopy appointment
2. 50-75 years of age
3. Due for CRC screening or surveillance (defined as no evidence of: colonoscopy in the past 5 years, fecal immunochemical testing in the past 12 months, flexible sigmoidoscopy or CT colonography in the past 5 years, stool DNA test or Cologuard in the last 3 years)

Exclusion Criteria:

1. Age <50 or >75
2. Pregnant woman
3. Evidence of prior colonoscopy in the past 5 years, fecal immunochemical testing in the past 12 months, flexible sigmoidoscopy or CT colonography in the past 5 years, fecal DNA test or Cologuard in the last 3 years
4. History of colorectal cancer
5. History of inflammatory bowel disease (Crohn's disease or Ulcerative colitis)
6. History of colon surgery or resection
7. History of symptoms concerning for colorectal cancer, such as lower GI bleeding, within the past 6 months
8. Family history of a hereditary colorectal cancer syndrome, such as familial adenomatous polyposis (FAP) or hereditary non-polyposis colon cancer (HNPCC)
9. Current serious medical condition with estimated life expectancy of less than 6 months, such as incurable cancer, end-stage congestive heart failure, decompensated cirrhosis, end stage renal disease, etc.
10. Dementia
11. Does not speak English
12. No telephone number listed in electronic medical record
13. Has any other condition that, in the opinion of the investigator, excludes the patient from participating in this study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Colonoscopy completion rate | 120 days
  The ratio of the number of participants who complete a colonoscopy to the total number of enrolled participants

SECONDARY OUTCOMES:
Colonoscopy scheduling rate | 120 days
  The ratio of the number of participants who schedule a colonoscopy to the total number of enrolled participants

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Kochman, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oyalowo A, Forde KA, Lamanna A, Kochman ML. Effect of Patient-Directed Messaging on Colorectal Cancer Screening: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e224529. doi: 10.1001/jamanetworkopen.2022.4529. PMID 35357457